CLINICAL TRIAL: NCT03581461
Title: Trauma-Informed Mindfulness-Based Yoga Intervention for Juvenile Justice-Involved Youth
Brief Title: Trauma-Informed Mindfulness-Based Yoga
Acronym: TIMBY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Kaiser Foundation Research Institute (Other); UConn Health (Other); New York University (Other)
Responsible Party: Principal Investigator, Ashli Owen-Smith, Assistant Professor, Georgia State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34AT009538 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-07-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Trauma
Keywords: Trauma; Yoga; Mindfulness
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-Informed Mindfulness-Based Yoga (Experimental): The TIMBY program will involve twice weekly, 1-hour long sessions that will incorporate the central elements of Hatha Yoga - breathwork (pranayama), physical postures (asana) and meditation.
  Interventions: Behavioral: Trauma-Informed Mindfulness-Based Yoga

INTERVENTIONS:
Behavioral: Trauma-Informed Mindfulness-Based Yoga — The TIMBY program will involve twice weekly, 1-hour long sessions that will incorporate the central elements of Hatha Yoga - breathwork (pranayama), physical postures (asana) and meditation.

SUMMARY:
The proposed study aims to gather the multiple types of preliminary data needed to design a large and rigorous pragmatic, cluster randomized trial on the impact of a trauma-informed mindfulness-based yoga program on enhancing self-regulation (in the short-term) and reducing recidivism (in the long-term) among juvenile justice-involved youth. Such a study will ultimately provide more definitive outcomes related to the effectiveness of these programs this population. If effective, the assimilation of such programs into the treatment plans of youth in juvenile justice facilities and in other residential settings could have a significant impact on a range of health, educational, vocational, and interpersonal outcomes relevant to this population.

DETAILED DESCRIPTION:
There are a number of interventions that aim to reduce recidivism among youth in the juvenile justice (JJ) system, some of which have documented evidence of effectiveness. However, the average reduction in recidivism following the implementation of these programs is modest at best, leaving a majority of JJ-involved youth at risk for recidivism. Many previous interventions have not been designed to address trauma-related symptoms despite evidence that most youth in the JJ system have a history of trauma and exposure to traumatic events is a predictor of recidivism. The pathway by which trauma exposure can lead to and perpetuate delinquency may be explained by some of the survival-oriented biological changes that occur in the brain of children who have been exposed to trauma - namely the compromised self-regulation systems that are responsible for reward/motivation, distress tolerance and executive function. As a result, youth with a history of trauma often have an impaired ability to modulate their behavioral and cognitive responses to a wide range of stressors. Thus, in light of the prevalence of trauma exposure in this population, interventions for JJ-involved youth should address trauma and, specifically, provide youth with resources related to enhancing self-regulation skills. Though some trauma-informed interventions have demonstrated empirical evidence of effectiveness with JJ-involved youth, many have methodological limitations and have not tested whether complementary mindfulness or somatically-oriented interventions can reduce recidivism by enhancing self-regulation in this population. The investigators propose to refine, implement and evaluate a trauma-informed, mindfulness-based yoga intervention that will enhance self-regulation among youth in the Georgia Department of Juvenile Justice (DJJ) system. The objectives of this mixed-methods investigation are to refine and pilot a trauma-informed, mindfulness-based yoga (TIMBY) program, assess the preliminary impact of this program on youth behavioral and psychosocial outcomes and test key aspects of the study design to inform the design of a full scale trial. The aims of this proposal are: (1) employ an iterative drafting and revision process to refine a trauma-informed yoga intervention specifically for youth in the JJ system, (2) conduct an initial pilot of the draft TIMBY intervention with JJ-involved youth at 2 DJJ facilities and (3) conduct and evaluate a small scale feasibility study of the TIMBY intervention. The expected products of the proposed research include a refined intervention protocol and manual of procedures, preliminary data regarding the impact of the intervention on participant outcomes, and data on intervention acceptability, adherence, fidelity, dose/duration, participant recruitment, retention and attrition, assessment feasibility and other barriers and facilitators to large-scale implementation. These products and data will enable a rapid launch of a subsequent, large-scale pragmatic cluster RCT funded through a future application.

ELIGIBILITY:
Inclusion Criteria:

* Detained at DeKalb Regional Youth Detention Center or the Atlanta Youth Development Campus (YDC)
* On the mental health caseload
* Male
* Ages 13-21
* English-speaking
* Able to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Recent (within the last week) serious non-compliant behavior (e.g., episodes of violent behavior requiring restraints or resulting in legal charges)
* Have current, untreated psychosis
* Are cognitively or decisionally impaired
* Are Wards of the State of Georgia

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in self-regulation as assessed by the Abbreviated Dysregulation Inventory (ADI) | Baseline and at 6- and 12-weeks follow-up
  The primary outcome of interest is changes in self-regulation, which will be assessed using the Abbreviated Dysregulation Inventory (ADI). The ADI is a 30-item self-report measure designed to assess 3 aspects of dysregulation - cognitive, emotional and behavioral - among adolescents. Each item on the ADI is rated on a four-point scale from 0 (never true) to 3 (always true).

SECONDARY OUTCOMES:
Changes in externalizing and internalizing behavior as assessed by The Child Behavior Checklist - Youth Self-Report (YSR). | Baseline and at 6- and 12-weeks follow-up
  Internalizing and externalizing behaviors will be measured using two subscales from The Child Behavior Checklist - Youth Self-Report (YSR). The YSR (18) is a self-report questionnaire divided in two parts: 1) Competencies and 2) Problems. It consists of 112 problem items covering different symptoms/behaviors each to be rated on a three-point scale (2 indicates that the symptom is present most of the time or applies well, 1 indicates that the symptom is present some of the time or applies to some extent, and 0 indicates the absence of symptom or problem behavior). All ratings refer to symptoms or problems experienced during the preceding 6 months.
Changes in anger as assessed by the State-Trait Anger Expression Inventory (STAXI-2) | Baseline and at 6- and 12-weeks follow-up
  Anger will be measured using the 57-item State-Trait Anger Expression Inventory (STAXI-2) which assesses youth's experience with and expression/control of anger. Specifically, the STAXI-2 includes self-report scales that measure State Anger, Trait Anger, Anger Expression-Out, Anger Expression-In, Anger Control-Out, Anger Control-In, and Anger Expression Index. Ratings are on a 4-point forced-choice response scale ("Not at all" to "Almost Always"). The State Anger scale measures transient anger intensity, while the Trait Anger scale measures the frequency of angry feelings. The Anger Expression-In scale measures the extent to which one "holds things in" or suppresses anger, whereas the Anger Expression-Out scale measures the actual expression of aggression. The Anger Control-In scale measures the extent to which the suppression of anger is controlled, whereas the Anger Control-Out scale measures the constraint of overt anger expression.
Changes in trauma-related symptoms as assessed by the Structured Trauma-Related Experiences and Symptoms Screener (STRESS) | Baseline and at 6- and 12-weeks follow-up
  Trauma-related symptoms will be assessed using the Structured Trauma-Related Experiences and Symptoms Screener (STRESS) which inventories 25 adverse childhood experiences/potentially traumatic events and assesses symptoms of PTSD. The STRESS assesses the four DSM-5 PTSD symptom clusters, dissociative symptoms, and trauma-related functional impairment (i.e., ability to make or keep friends, get along with other kids, do schoolwork, get along with teachers, get along with household, and get chores done) using 21 items measured on a 4-point rating scale (none, 1 day, 2-3 days, and most days). The STRESS uses a briefer retrospective time frame when assessing symptoms based on evidence that children's retrospective report is less valid over an extended period of time (De Los Reyes & Kazdin, 2005).
Changes in impulsivity as assessed by the Barratt Impulsiveness Scale (BIS) | Baseline and at 6- and 12-weeks follow-up
  Impulsivity will be assessed using the Barratt Impulsiveness Scale (BIS), which is a 30-item 4-point rating scale ("rarely/never" to "almost always/always") and captures 3 domains of impulsivity: cognitive impulsiveness which involves making quick decisions (e.g., "I make up my mind quickly"), motor impulsiveness which involves acting without thinking (e.g., "I act on the spur of the moment"), and non-planning impulsiveness which involve a lack of ''futuring" or forethought (e.g., "I am more interested in the present than the future").
Changes in psychological flexibility as assessed by the Acceptance and Action Questionnaire (AAQ-II) | Baseline and at 6- and 12-weeks follow-up
  Psychological flexibility will be assessed using the Acceptance and Action Questionnaire (AAQ-II) is the most widely used measure of experiential avoidance and psychological inflexibility. The AAQ-II is a seven-item self-report measure that uses a 7-point Likert scale (1=never true, 7=always true). Sample items include "I am afraid of my feelings" and "Emotions cause problems in my life." Three of the AAQ-II items are taken directly from the nine-item AAQ.
Changes in mindfulness as assessed by the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | Baseline and at 6- and 12-weeks follow-up
  Mindfulness will be assessed using the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a 12-item measure designed to measure four core characteristics of mindfulness described by Kabat-Zinn (1990): (1) the ability to regulate attention ["I have a hard time concentrating on what I am doing," (reverse-scored)], (2) an orientation to present or immediate experience [e.g., "I focus on the present moment", "I am preoccupied with the past" (reverse scored)], (3) awareness of experience (e.g., "It's easy for me to keep track of my thoughts and feelings"), and (4) an attitude of acceptance or nonjudgment towards experience (e.g., "I believe it is OK to be sad or angry"). Participants respond on a 4-point Likert scale from "Rarely/not at all" to "Almost always."

CONTACTS AND LOCATIONS:
Overall Officials: Ashli Owen-Smith, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No